CLINICAL TRIAL: NCT00973271
Title: A Multi-Center, Randomized, Double-Blind, Placebo- and Active-Controlled Study Assessing the Efficacy, Safety and Tolerability of Diazoxide Choline Controlled-Release Tablet (DCCR) in Subjects Without Diabetes Mellitus Having Very High Fasting Triglyceride Levels, With Double-Blind Active-Controlled Extension Assessing Safety and Tolerability
Brief Title: Diazoxide Choline Controlled-Release Tablet (DCCR) for Very High Triglycerides
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Did not continue with development of DCCR in Very High Triglycerides
Sponsor: Essentialis, Inc. (Industry)
Responsible Party: Neil M. Cowen, PhD, Chief Scientific Officer, Essentialis, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PV011
Record Dates: First submitted 2009-09-05; First posted 2009-09-09 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Hypertriglyceridemia
Keywords: hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia | interventions — fenofibric acid; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 290 mg DCCR (Experimental)
  Interventions: Drug: 290 mg DCCR; Drug: Placebo; Drug: atorvastatin
- 435 mg DCCR (Experimental)
  Interventions: Drug: 435 mg DCCR; Drug: Placebo; Drug: atorvastatin
- 135 mg fenobric acid (Active Comparator)
  Interventions: Drug: 135 mg fenofibric acid; Drug: Placebo; Drug: atorvastatin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: atorvastatin

INTERVENTIONS:
Drug: 290 mg DCCR — 290 mg diazoxide choline
  Arms: 290 mg DCCR
Drug: 435 mg DCCR — 435 mg diazoxide choline
  Arms: 435 mg DCCR
Drug: 135 mg fenofibric acid — 135 mg fenofibric acid
  Other Names: 135 mg fenobric acid
  Arms: 135 mg fenobric acid
Drug: Placebo — Placebos matching each of 2 doses of DCCR and 135 mg fenofibric acid
  Other Names: Placebos matching DCCR and fenofibric acid
Drug: atorvastatin — 20 mg atorvastatin
  Other Names: 20 mg atorvastatin

SUMMARY:
The hypothesis of this study is that DCCR is effective as both monotherapy and in combination with a statin in lowering triglycerides in subjects with very high triglycerides

DETAILED DESCRIPTION:
Very high triglyceride is a risk for pancreatitis. Studies have shown Diazoxide Choline has the potential to effectively lower triglycerides in patients with very high triglycerides.

ELIGIBILITY:
INCLUSION CRITERIA:

Fasting triglycerides

* Difference between Visit 3 (7 days prior to Baseline Visit) and Visit 4 (3 days prior to Baseline Visit) ≤ 60% (compared to the higher value of Visit 3 or Visit 4)
* Run-in Triglycerides* ≥ 500 mg/dL and < 1500 mg/dL *Run-in Triglyceride is defined as the average fasting triglycerides for Visit 3 (7 days prior to Baseline Visit) and Visit 4 (3 days prior to Baseline Visit).

Statin use

* Either Statin-naive

  - Must not be on statin at Screening and remaining as such during the Run-in/Washout Period and throughout the study
* Or Statin-treated

  * Must be receiving a stable and effective dose of statin for ≥ 3 months without significant side effects or intolerance prior to Screening
  * Must be willing to switch to 20 mg atorvastatin at the start of the Run-in/Washout Period and continue throughout the study

Medication washout

* All subjects must be willing to undergo washout of all other lipid-lowering medications

Fasting LDL cholesterol

* ≤ l60 mg/dL at both Screening Visit and Visit 4

Glycemic status

* Fasting glucose < 126 mg/dL at Screening Visit
* HbA1c < 6.5% at Screening Visit

EXCLUSION CRITERIA:

Medications: recent, current, anticipated

* Administration of investigational drugs within 1 month prior to Screening Visit
* Thyroid hormones or preparations within 1 month prior to Screening Visit (except in subjects on stable dose of replacement therapy for at least 1 month)
* Thiazide diuretics within 2 weeks prior to Screening Visit
* Discontinuation of beta-blockers within 1 month prior to Screening Visit or planned discontinuation of beta-blocker therapy
* Anticipated requirement for use of prohibited concomitant medications

History of allergic reaction or significant intolerance to:

* Diazoxide
* Thiazides
* Sulfonamides
* Fenofibrate or fenofibric acid derivatives

Lifestyle changes

• Subjects intending to change exercise habits, quit smoking and/or quit alcohol use during the initial 12-week Placebo-Controlled Treatment Period of the study

Specific diagnoses, medical conditions and history

* Known type I or III hyperlipidemia
* Known type 1 DM
* Known type 2 DM
* Any other clinically significant endocrine, cardiovascular, pulmonary, neurological, psychiatric, hepatic, gastrointestinal, hematological, renal, or dermatological disease interfering with the assessments of the study medications, according to the Investigator

Specific laboratory test results

• Any relevant biochemical abnormality interfering with the assessments of the study medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-03; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The effect of DCCR on triglycerides in subjects without diabetes mellitus who have very high triglycerides over a period of 84 days | 84 days

SECONDARY OUTCOMES:
The effects of DCCR on Apo B and non-HDL in subjects without diabetes mellitus who have very high triglycerides over a period of 84 days | 84 days